CLINICAL TRIAL: NCT00998049
Title: Phase II Trial of Intravenously Administered AMD3100 (Plerixafor) for Stem Cell Mobilization in Patients With Multiple Myeloma Undergoing Autologous Stem Cell Transplantation Following a Lenalidomide Based Initial Therapy
Brief Title: Plerixafor in Treating Patients With Multiple Myeloma Previously Treated With Lenalidomide and Planning to Undergo Autologous Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0889; NCI-2009-01328 (Registry Identifier: NCI-CTRP); MC0889 (Other: Mayo Clinic Cancer Center); 08-005644 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma; Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plerixafor (Experimental): Plerixafor 160mg/kg/dose by IV on days 5-8
  Filgrastim (G-CSF) 10 mg/kg/dose subcutaneously on days 1-8.
  Interventions: Drug: plerixafor; Drug: filgrastim

INTERVENTIONS:
Drug: plerixafor — Plerixafor 160mg/kg/dose by IV on days 5-8
  Other Names: AMD 3100; LM-3100; Mozobil
Drug: filgrastim — Filgrastim (G-CSF) 10 mg/kg/dose subcutaneously on days 1-8.
  Other Names: G-CSF; granulocyte colony-stimulating factor; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor

SUMMARY:
Rationale: Giving colony-stimulating factors, such as G-CSF and plerixafor helps stem cells move from the patient's bone marrow to the blood so they can be collected and stored. Purpose: This phase II trial is studying how well plerixafor works in patients with multiple myeloma previously treated with lenalidomide and planning to undergo autologous stem cell transplant.

DETAILED DESCRIPTION:
Primary Objective: I. To determine the proportion of patients reaching a stem cell yield of 3 million CD34 cells/kg by second day of apheresis with intravenously administered AMD3100 among patients receiving primary therapy for myeloma with lenalidomide. Secondary Objectives: I. Safety and tolerability of intravenously administered AMD3100. II. Rate of failure to mobilize. Outline: Patients receive plerixafor IV on days 5-8 and filgrastim subcutaneously on days 1-8 in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
Inclusion - Absolute neutrophil count >= 1000/uL - Platelet >= 75000/uL - Hemoglobin >= 8.0 g/dL - Serum aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT), serum alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) and total bilirubin < 2 x upper limit of normal (ULN) - Confirmed diagnosis of multiple myeloma, requiring therapy - Initial treatment for symptomatic myeloma using a lenalidomide based treatment regimen, started =< 12 months prior to registration - Received at least 2 cycles of treatment with the lenalidomide regimen - Last dose of lenalidomide > 2 weeks prior to registration - Eligible to undergo autologous transplantation - ECOG performance status (PS) 0 or 1 - Willingness to return for follow-up - Provide informed written consent - Adequate cardiopulmonary function: ejection fraction >= 45%, corrected pulmonary diffusion capacity of >= 50%, FEV1 >= 50%, FVC >= 50% - Negative serum or urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only Exclusion - A co-morbid condition which, in the view of the Investigators, renders the patient at high risk from treatment complications - Active malignancy with the exception of non melanoma skin cancer or in situ cervical or breast cancer - Other co-morbidity which would interfere with patient's ability to participate in the trial, e.g. uncontrolled infection, uncompensated heart or lung disease - Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational - Use of cyclophosphamide as part of stem cell mobilization - Use of more than one regimen for treatment of symptomatic myeloma - Dialysis dependent renal failure - Pregnant women or women of reproductive ability who are unwilling to use effective contraception - Nursing women - Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment - Acute infection, active HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, M.D., Study Chair — Mayo Clinic; Joseph R. Mikhael, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty (40) participants were recruited at Mayo Clinic (Rochester, Florida and Arizona) between December 2009 and October 2011.
Pre-assignment Details: One participant was deemed ineligible and is excluded from all analyses per study design.
Period: Overall Study
Arm/Group | Plerixafor
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Plerixafor
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 60 [28 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving 3 Million CD34 Cells/kg After 2 Days of Apheresis
Description: Number of CD34 cells/kg collected on days 1-2.
  Apheresis is the process when blood is taken out through a catheter in a vein in one arm, blood is sent through a machine that takes out the stem cells and the rest of the blood is then returned through a vein in your other arm.
Time Frame: After 2 days of apheresis
Measure: Number; unit: participants
Arm/Group | Plerixafor
Number analyzed (Participants) | 39
participants | 38

2. Secondary Outcome: CD34 Yield on Day 1
Description: Number of CD34 cells/kg collected on day 1.
Time Frame: Day 1
Measure: Median (Full Range); unit: cells/kg
Arm/Group | Plerixafor
Number analyzed (Participants) | 39
cells/kg | 3870000 [670000 to 9160000]

3. Secondary Outcome: CD34 Yield Day 2
Description: Number of CD34 cells/kg collected on day 2
Time Frame: Day 2
Measure: Median (Full Range); unit: cells/kg
Arm/Group | Plerixafor
Number analyzed (Participants) | 39
cells/kg | 3550000 [470000 to 9170000]

4. Secondary Outcome: Median Number of Days of Apheresis
Time Frame: Duration of apheresis (up to 7 days)
Measure: Median (Full Range); unit: days
Arm/Group | Plerixafor
Number analyzed (Participants) | 39
days | 4 [2 to 5]

5. Secondary Outcome: Time to Reach 6 Million CD34 Cells
Description: Number (median and 95% confidence interval) of days to reach 6 million CD34 cells/kg was estimated using the Kaplan Meier method. Participants were lower than 6 million CD34 cells/kg at time of last follow-up will be censored at that date.
Time Frame: Duration of apheresis (up to 7 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Plerixafor
Number analyzed (Participants) | 39
days | 5 [5 to 6]

6. Secondary Outcome: Rate of Failure to Mobilize
Description: The rate of failure to mobilize will be estimated by dividing the number of patients that fail to mobilize by the total number of evaluable patients. A patient is considered a failure if they never achieve 2.5 million CD34 cells/kg.
Time Frame: Duration of apheresis (up to 7 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plerixafor
Number analyzed (Participants) | 39
percentage of participants | 3 [.006 to 13]

ADVERSE EVENTS:
Arm/Group | Plerixafor
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 25/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plerixafor (N=39)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Bloating (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 17 (17)
Injection site reaction (General disorders) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes